CLINICAL TRIAL: NCT06741813
Title: Allogeneic Versus Autologous Hematopoietic Stem Cell Transplantation for Adult T Lymphoblastic Lymphoma as First-line Consolidation.
Brief Title: Allo-HSCT vs ASCT in Adult T-LBL
Acronym: TROPHY-NHL01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peking University People's Hos
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: T Lymphoblastic Lymphoma
Keywords: allogeneic hematopoietic stem cell transplantation; Autologous hematopoietic stem cell transplantation; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: For the adult patients (≥ 18 years) with Ann-Arbor stage III or IV T-LBL and achieving CR after 3 courses of induction chemotherapy, all the patients who fulfilled inclusion/exclusion criteria were randomly assigned in a 1:1 ratio to receive ASCT (ASCT group) or receive allo-HSCT (Allo-HSCT group). Patients would receive additional 1 course of chemotherapy after randomization and then received HSCT. Then we compared the clinical outcomes between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASCT group (Active Comparator): T-LBL patients achieving CR after induction chemotherapy and then received ASCT as first line consolidation
  Interventions: Procedure: ASCT
- Allo-HSCT (Experimental): T-LBL patients achieving CR after induction chemotherapy and received allo-HSCT as first line consolidation
  Interventions: Procedure: Allo-HSCT

INTERVENTIONS:
Procedure: ASCT — The chemotherapy-based preconditioning regimen was BeEAM, which consisted of bendamustine (120-180 mg·m-2·day-1，days -8 to -7), etoposide (200 mg·m-2·day-1，days -6 to -3), cytarabine (400 mg·m-2·day-1，days -6 to -3), and melphalan (140 mg·m-2·day-1，days -2).
  Arms: ASCT group
Procedure: Allo-HSCT — Chemotherapy-based preconditioning regimen consisted of cytarabine 4 g·m-2·day-1 (days -9), busulfan (3.2 mg·kg-1·day-1 administered intravenously on days -8 to -6) (day 0 being the first day of donor cell infusion), cyclophosphamide (1.8 g·m-2·day-1, days -5 to -4), and semustine (250 mg.m-2, day -3). For the patients older than 55 years old or with HCT-CI score of 3 or more, cyclophosphamide can be decreased to 1.0 g·m-2·day-1, days -5 to -4, and added fludarabine (30mg·m-2·day-1, days -6 to -2). Rabbit antithymocyte globulin (thymoglobulin, 1.5 to 2.5 mg/kg, days -5 to -2; Sanofi, France) was administered to the HID and URD groups or MSD HSCT recipients who older than 40 years old (1.5 mg/kg, days -4 to -2).
  All MSD, HID, and URD HSCT recipinets received cyclosporine A (CsA), mycophenolate mofetil (MMF), and short-term methotrexate (MTX) for GVHD prophylaxis. CsA (2.5 mg/kg, q12h, intravenous [i.v.]) was used from day -9, of which the trough concentration was adjusted to 150-250 ng
  Arms: Allo-HSCT

SUMMARY:
Autologous hematopoietic stem cell transplantation (ASCT) is the important consolidation for adult T-LBL. Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is also the important consolidation for adult T-LBL. So ASCT vs allo-HSCT: which is better consolidation for adult T-LBL?

DETAILED DESCRIPTION:
1. Characteristics of adult T-lymphoblastic lymphoma (T-LBL) T-lymphoblastic lymphoma (T-LBL) is a highly aggressive lymphoma which shares biological and morphological features with T-cell acute lymphoblastic leukemia (T-ALL), and T-LBL is conventionally distinguished from T-ALL by less than 25% bone marrow (BM) infiltrating blasts cells. T-LBL only represents 3-4% of adult's non-Hodgkin lymphomas (NHL) which is a rare histologic subtype of NHL in adults. For this reason, few studies had focused on the disease-specific cohort of adult T-LBL patients and most of the studies included both T-LBL and T-ALL.
2. Autologous hematopoietic stem cell transplantation (ASCT) is the important consolidation for adult T-LBL The treatment paradigm of T-LBL is evolving. In the 1980s, when patients were treated with lymphoma-like regimens, the outcome of T-LBL was dismal and the 5-year progression-free survival (PFS) and overall survival (OS) was only 22% and 32%, respectively. ALL-like regimens significantly increase the complete response (CR) rate to more than 90% in T-LBL patients; however, disease relapse negatively impacts the long-term survival. For example, the 3-year OS rates of T-LBL could be as high as 66.9% to 70% while the 5-year OS rates decrease to below 50% in adults.

   ASCT is an important consolidation for adult T-LBL, which could also improve the survival of T-LBL compared with those only receiving chemotherapy. However, for patients with some risk factors (such as central nervous system [CNS] involvement or bone marrow [BM] involvement), the survival was very poor. In addition, ASCT is associated with a significantly higher risk of disease progression or recurrence.
3. Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is also the important consolidation for adult T-LBL Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is one of the most important curative treatments for T-LBL mainly because of the graft-versus-lymphoma effect, particularly for those with high-risk characteristics of relapse. Recently, in a multicenter study of China enrolled 130 Ann-Arbor stage III or IV T-LBL patients (> 16 years) treated with allo-HSCT, the 2-year probabilities of disease progression, PFS, OS and NRM after allo-HSCT were 21.0%, 69.8%, 79.5%, and 9.2%, respectively. Patients with CNS involvement had a higher cumulative incidence of disease progression compared with those without CNS involvement (57.1% vs. 18.9%, P = 0.014). Patients receiving allo-HSCT in non-remission (NR) had a poorer PFS compared with those receiving allo-HSCT in complete remission (CR) or partial remission (PR) (49.2% vs. 72.7%, P = 0.041). Particularly, for patients with BM involvement and achieving CR before allo-HSCT, measurable residual disease (MRD) positivity before allo-HSCT was associated with a poorer PFS compared with MRD negativity (62.7% vs. 86.8 %, HR 1.94, P = 0.036). Thus, this real-world data suggested that allo-HSCT appeared to be an effective therapy for adults T-LBL patients with Ann-Arbor stage III or IV disease.
4. ASCT vs allo-HSCT: which is better consolidation for adult T-LBL Thus far, whether allo-HSCT could be superior to ASCT as consolidation in T-LBL was unknown, which should be identified by randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* 1) Newly diagnosed T-LBL; 2) 18-65 years of age at the time of diagnosis; 3) Categorized into Ann-Arbor stage III or IV; 4) Achieving complete response (CR) after 3 courses of induction chemotherapies; 5) ECOG PS score 0 or 1; 6) It needs consent from the patients or/and legal guardian, and signature on the Informed Consent.

Exclusion Criteria:

* 1) Newly diagnosed T-LBL, but categorized into Ann-Arbor stage I or II; 2) < 18 years, or older than 65 years at the time of diagnosis; 3) Achieving CR after 4 or more courses of induction chemotherapies, or could not achieve at least CR after induction chemotherapies; 4) with > 25% BM involvement or > 5% lymphoma cells in the peripheral blood; 5) ECOG PS score of 2 or more; 6) Patients with other comorbidities or mental diseases that influence the life safety and compliance of patients as well as affect informed consent, enrollment in the research, follow-up visit or result interpretation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Probability of PFS at months 1, 2, 6, 12, 18 & 24 will be estimated from the Kaplan-Meier curves for each arm.
  Progression-free survival (PFS), defined as the time from the date of randomization to the date of disease progression/relapse, or death due to any cause.

SECONDARY OUTCOMES:
Relapse | Cumulative incidence of disease progression/relapse at months 1, 2, 6, 12, 18 & 24 will be estimated, considering non-relapse mortality as competing events.
  Relapse, defined as the time from date of randomization to date of disease progression/relapse.
Non-relapse mortality (NRM) | Cumulative incidence of NRM at months 1, 2, 6, 12, 18 & 24 will be estimated, considering disease progression/relapse as competing events.
  NRM, defined as the time from date of randomization to date of death not preceded by disease progression/relapse.
Overall survival (OS) | Probability of overall survival at months 1, 2, 6, 12, 18 & 24 will be estimated from the Kaplan-Meier curves for each arm.
  OS, defined as the time from the date of randomization to the date of death due to any cause.

IPD SHARING:
Plan to Share IPD: No